CLINICAL TRIAL: NCT00006219
Title: A Phase II Clinical Trial of Dehydroepiandrosterone and Biaxin in Monoclonal Gammopathy of Undetermined and Borderline Significance
Brief Title: Chemoprevention Therapy in Treating Patients at High Risk of Developing Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: John A. Lust, M.D., Mayo Clinic Cancer Center
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000068084; P30CA015083 (NIH); 979202 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Clarithromycin; Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: clarithromycin
Drug: prasterone

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. Dehydroepiandrosterone and clarithromycin may be effective in preventing multiple myeloma.

PURPOSE: Randomized phase II trial to compare the effectiveness of dehydroepiandrosterone with that of clarithromycin in treating patients who may be at a high risk of developing multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether dehydroepiandrosterone (DHEA) or clarithromycin causes a significant reduction in bone marrow plasmacytosis, serum and/or urine M protein or Bence Jones protein, and surrogate endpoint biomarkers in patients with monoclonal gammopathy of undetermined or borderline significance.
* Determine whether differences in interleukin-1-beta (IL-1-beta) expression and IL-1-beta dependent biomarkers (adhesion molecule expression and serum interleukin-6 levels) are useful surrogate endpoint biomarkers in these patients.
* Determine whether differences in ploidy, proliferative index, nuclear pleomorphism index, circulating monoclonal plasma cells, Th1/Th2 ratios, serum s-interleukin-6R (SIL-6R) levels, interleukin-6 and SIL-6R expression, or plasma cell apoptosis assay are useful surrogate endpoint biomarkers in these patients.
* Determine the effects of these treatment regimens on the quality of life of these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to disease (monoclonal gammopathy of undetermined significance vs monoclonal gammopathy of borderline significance) and monoclonal protein abnormality (IgG vs IgA). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive oral dehydroepiandrosterone (DHEA) once daily.
* Arm II: Patients receive oral clarithromycin once or twice daily.
* Arm III: Patients receive oral placebo once daily.
* Arm IV: Patients receive oral placebo twice daily. Treatment continues for 6 months in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, 6 months, 12 months, and then at disease progression.

Patients are followed every 3 months for 1 year and then every 6 months for 1.5 years.

PROJECTED ACCRUAL: A total of 75 patients (25 per treatment arms I and II and 25 between arms III and IV) will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* New or prior diagnosis of 1 of the following:

  * Monoclonal gammopathy of undetermined significance

    * Bone marrow plasma cells of less than 10%
  * Monoclonal gammopathy of borderline significance

    * Bone marrow plasma cells of 10-30%
* Serum IgG or IgA at least 1.5 g/dL
* Bone marrow plasmacytosis no greater than 30%
* No multiple myeloma, amyloidosis, or B-cell neoplasm
* No evidence of bone lesions
* Prostate-specific antigen less than 4 ng/mL

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN) (unless history of Gilbert's disease)
* AST and ALT no greater than 1.5 times ULN (unless history of Gilbert's disease)

Renal:

* Creatinine no greater than 1.8 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No prior thromboembolic event within the past 5 years

Other:

* No prostate cancer or clinically significant benign prostatic hypertrophy
* No prior malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No malignancy suspected on mammogram
* No hypersensitivity to DHEA, clarithromycin, or any macrolide antibiotic (e.g., erythromycin)
* No insulin-dependent diabetes
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier method of contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* At least 30 days since prior DHEA or other steroids that may affect M protein

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 30 days since prior clarithromycin
* At least 30 days since any other prior agents that may affect M protein
* No concurrent cisapride, terfenadine, pimozide, astemizole, or loratadine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A. Lust, MD, PhD, Study Chair — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota